CLINICAL TRIAL: NCT06028685
Title: Acupoint Stimulation Improves Fatigue and Sleep Quality in Patients With Postdialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-06-002B
Record Dates: First submitted 2023-07-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Hemodialysis
Keywords: fatigue; sleep
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: This study adopts an experimental research design.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study employs computer-based random allocation, where the assignments are sealed in opaque envelopes. The researchers open the envelopes to distribute participants into the experimental and control groups, ensuring blinding of the study participants. The data analysts responsible for statistical analysis are separate individuals who are unaware of the participants' grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): The experimental group will receive low-level laser stimulation on seven acupoints. The stimulation will be administered three times per week for a duration of six weeks.
  Interventions: Device: Acupoint stimulation
- control group (Placebo Comparator): The control group will receive sham low-level laser stimulation on the acupoints, without emitting laser beams.
  Interventions: Device: Acupoint stimulation(placebo)

INTERVENTIONS:
Device: Acupoint stimulation — The experimental group will receive low-level laser stimulation on seven acupoints, including Shenmen (HT7), Neiguan (PC6), Hegu (LI4), Zusanli (ST36), Yanglingquan (GB34), Sanyinjiao (SP6), and Taixi (KI3). The stimulation will be administered three times per week for a duration of six weeks.
  Arms: experimental group
Device: Acupoint stimulation(placebo) — The control group will receive sham low-level laser stimulation on seven acupoints, including Shenmen (HT7), Neiguan (PC6), Hegu (LI4), Zusanli (ST36), Yanglingquan (GB34), Sanyinjiao (SP6), and Taixi (KI3), without emitting laser beams.The stimulation will be administered three times per week for a duration of six weeks.
  Arms: control group

SUMMARY:
Hemodialysis is a necessary treatment to prolong the lives of patients with end-stage kidney disease. However, long-term dialysis can lead to fatigue and decreased sleep quality. Acupoint stimulation can regulate meridians and improve physical function. Nevertheless, the effectiveness of low-level laser stimulation on fatigue and sleep quality in hemodialysis patients remains unclear.

This study is designed to use low-level laser stimulation as an intervention measure to evaluate its effectiveness in improving fatigue and sleep quality in hemodialysis patients.

DETAILED DESCRIPTION:
Hemodialysis is a necessary treatment to prolong the lives of patients with end-stage kidney disease. However, long-term dialysis can lead to fatigue and decreased sleep quality. Acupoint stimulation can regulate meridians and improve physical function. Nevertheless, the effectiveness of low-level laser stimulation on fatigue and sleep quality in hemodialysis patients remains unclear.

This study is designed to use low-level laser stimulation as an intervention measure to evaluate its effectiveness in improving fatigue and sleep quality in hemodialysis patients.

The experimental group will receive low-level laser stimulation on seven acupoints, including Shenmen (HT7), Neiguan (PC6), Hegu (LI4), Zusanli (ST36), Yanglingquan (GB34), Sanyinjiao (SP6), and Taixi (KI3). The stimulation will be administered three times per week for a duration of six weeks. The control group will receive sham low-level laser stimulation on the acupoints, without emitting laser beams.

Before and after each intervention, fatigue will be measured using a visual analog scale for a total of 18 measurements. Additionally, at baseline and at the 2nd, 4th, and 6th weeks, the hemodialysis patients will be assessed using the Fatigue Scale for Hemodialysis Patients, Dialysis Recovery Time Scale, Pittsburgh Sleep Quality Index, Dialysis Symptom Index, and Beck Depression Inventory.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20 years and above.
2. Diagnosed with end-stage kidney disease and receiving regular outpatient hemodialysis three times a week for at least three months.
3. Conscious and capable of communication in Mandarin or Taiwanese (Hokkien).
4. Willing to participate in this study and have signed the informed consent form.

Exclusion Criteria:

1. Presence of skin lesions or infectious wounds at the acupoint locations.
2. Taking immunosuppressive medication.
3. Photosensitivity or sensitivity to light.
4. Individuals with implanted cardiac pacemakers.
5. Patients using sleep medication.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
fatigue1 | Three times per week, for six weeks, totaling 18 sessions.
  The fatigue visual analogue scale：The score ranges from 0 to 10 points, with higher scores indicating a higher level of fatigue.
fatigue2 | measured at baseline and at the 2nd, 4th, and 6th weeks.
  Fatigue Scale for Hemodialysis Patients：The score ranges from 26 to 104 points, with higher scores indicating a higher level of fatigue.
fatigue3 | measured at baseline and at the 2nd, 4th, and 6th weeks.
  Dialysis recovery time: The recovery time is divided into four intervals, including less than 2 hours, 2-6 hours, 7-12 hours, and greater than 12 hours. This is determined by responses from dialysis patients regarding the time needed for recovery during dialysis treatment.
sleep | measured at baseline and at the 2nd, 4th, and 6th weeks.
  Pittsburgh Sleep Quality Index：The total score ranges from 0 to 21 points, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Rou-Yu Sung, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Sung RY, Yeh ML, Chen FP, Lo MY, Yu J. Laser acupuncture improves post-dialysis fatigue and sleep quality independent of time-varying dialysis and depression symptoms: a double-blind, randomized, placebo-controlled trial. BMC Complement Med Ther. 2025 Dec 13. doi: 10.1186/s12906-025-05203-3. Online ahead of print. PMID 41390393